CLINICAL TRIAL: NCT04333329
Title: Transcranial Pulse Stimulation for Alzheimer's Disease in an Open Prospective Pilot Study
Brief Title: Transcranial Pulse Stimulation (TPS) for Alzheimer's Disease (AD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Storz Medical AG (Industry)
Collaborators: Rheintalklinik (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU_14_032
Record Dates: First submitted 2018-09-06; First posted 2020-04-03 (Actual); Last update posted 2020-04-03 (Actual); Status verified 2020-04

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AD Patients (Experimental): All patients were treated with the TPS device (new name: NEUROLITH (Storz Medical AG))
  - 6 sessions within 2 weeks, each sessions consisting of 6000 TPS pulses of 0.2 mJ/mm²
  Interventions: Device: NEUROLITH

INTERVENTIONS:
Device: NEUROLITH — transcranial pulse stimulation (TPS)
  Other Names: transcranial pulse stimulation (TPS)

SUMMARY:
This is a prospective open comprehensive proof-of-principle pilot study.

DETAILED DESCRIPTION:
This is a prospective open comprehensive proof-of-principle pilot study with patients of mild to moderate Alzheimer's Disease who have been treated with transcranial pulse stimulation (TPS)

ELIGIBILITY:
Inclusion Criteria:

* Clinically stable patients with probable Alzheimer's Disease (Diagnosis according to ICD-10 Criteria (F00))
* MMSE ≥ 10: Mild and moderate Alzheimer's Disease according to AWMF Register, S3 Guidelines of DGN 038/013 and DEGAM 035/021
* At least 3 months of stable antidementia therapy or no antidementia therapy necessary (Patients need to continue their standard treatment within the clinical investigation according to the guidelines as TPS is considered an additional treatment to standard therapy)
* Signed written informed consent
* 18 years ≤ Age ≤ 85 years
* Monthly pregnancy tests for female patients in childbearing age

Exclusion Criteria:

* Non-compliance with the protocol (including CERAD-plus)
* Pregnancy
* Breast-feeding women
* Microbubbles (contrast agents) in application area
* Cerebral pathology unrelated to Alzheimer's disease
* Metallic objects in the head
* Neurosurgical intervention of the brain / Craniotomy
* Cardiac disorders
* History of psychiatric diseases before development of dementia
* Hemophilia or other blood clotting disorders
* Cortisone treatment up to 6 months before first treatment
* Other conditions implying increased risk according to the judgement of the investigator

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-08-08 (Actual); Primary Completion 2017-02-15 (Actual); Study Completion 2017-02-15 (Actual)

PRIMARY OUTCOMES:
Consortium to Establish a Registry for Alzheimer's Disease (CERAD) - Total Score | 3 months after treatment
  CERAD is a cognitive test battery which is normalized for age, gender and education. The CERAD total score ranges from 0 to 100 with 100 meaning "normal cognitive ability" and 0 meaning "severe cognitive impairment".
Adverse Device Effects | within 3 months follow-up
  Number of ADEs

SECONDARY OUTCOMES:
Consortium to Establish a Registry for Alzheimer's Disease (CERAD) - Total Score | Immediately post treatment (at 2 weeks)
  CERAD is a cognitive test battery which is normalized for age, gender and education. The CERAD total score ranges from 0 to 100 with 100 meaning "normal cognitive ability" and 0 meaning "severe cognitive impairment".
Consortium to Establish a Registry for Alzheimer's Disease (CERAD) - Total Score | 1 month after treatment (at 6 weeks)
  CERAD is a cognitive test battery which is normalized for age, gender and education. The CERAD total score ranges from 0 to 100 with 100 meaning "normal cognitive ability" and 0 meaning "severe cognitive impairment".
Mini-Mental-State Examination (MMSE) | Immediately post treatment (at 2 weeks)
  The MMSE consists of 10 items that cover orientation, short term memory, attentional capabilities, arithmetic performance and language functions. Scoring is possible between 0 (worst) and 30 (best).
Mini-Mental-State Examination (MMSE) | 1 month after treatment (at 6 weeks)
  The MMSE consists of 10 items that cover orientation, short term memory, attentional capabilities, arithmetic performance and language functions. Scoring is possible between 0 (worst) and 30 (best).
Mini-Mental-State Examination (MMSE) | 3 months after treatment (at 14 weeks)
  The MMSE consists of 10 items that cover orientation, short term memory, attentional capabilities, arithmetic performance and language functions. Scoring is possible between 0 (worst) and 30 (best).
Clock Drawing Test (CDT) | Immediately post treatment (at 2 weeks)
  The clock drawing test is used to assess visuoconstruction abilities. The subject is asked to draw the face of a clock with all numbers and to set the hands for a specified time (hh:mm). Scores range from 0 (worst) to 7 (best).
Clock Drawing Test (CDT) | 1 month after treatment (at 6 weeks)
  The clock drawing test is used to assess visuoconstruction abilities. The subject is asked to draw the face of a clock with all numbers and to set the hands for a specified time (hh:mm). Scores range from 0 (worst) to 7 (best).
Clock Drawing Test (CDT) | 3 months after treatment (at 14 weeks)
  The clock drawing test is used to assess visuoconstruction abilities. The subject is asked to draw the face of a clock with all numbers and to set the hands for a specified time (hh:mm). Scores range from 0 (worst) to 7 (best).
Beck Depression Inventory (BDI) | Immediately post treatment (at 2 weeks)
  The BDI measures the severity of depression. It is a 21-item questionnaire for self-evaluation with 0-3 scores per item. The total score is the sum of all items. It ranges from 0 (normal state) to 63 (severe depression).
Beck Depression Inventory (BDI) | 1 month after treatment (at 6 weeks)
  The BDI measures the severity of depression. It is a 21-item questionnaire for self-evaluation with 0-3 scores per item. The total score is the sum of all items. It ranges from 0 (normal state) to 63 (severe depression).
Beck Depression Inventory (BDI) | 3 months after treatment (at 14 weeks)
  The BDI measures the severity of depression. It is a 21-item questionnaire for self-evaluation with 0-3 scores per item. The total score is the sum of all items. It ranges from 0 (normal state) to 63 (severe depression).
Geriatric Depression Scale - short form (GDS-15) | Immediately post treatment (at 2 weeks)
  The Geriatric Depression Scale (GDS) is a questionnaire to assess depression in the elderly population. This scale generates self-evaluation scores concerning various aspects with relevance for the depressive disease (e.g. mood, drive, anxiety). The short form contains 15 items. The GDS-15 score ranges from 0 (normal state) to 15 (severe depression).
Geriatric Depression Scale - short form (GDS-15) | 1 month after treatment (at 6 weeks)
  The Geriatric Depression Scale (GDS) is a questionnaire to assess depression in the elderly population. This scale generates self-evaluation scores concerning various aspects with relevance for the depressive disease (e.g. mood, drive, anxiety). The short form contains 15 items. The GDS-15 score ranges from 0 (normal state) to 15 (severe depression).
Geriatric Depression Scale - short form (GDS-15) | 3 months after treatment (at 14 weeks)
  The Geriatric Depression Scale (GDS) is a questionnaire to assess depression in the elderly population. This scale generates self-evaluation scores concerning various aspects with relevance for the depressive disease (e.g. mood, drive, anxiety). The short form contains 15 items. The GDS-15 score ranges from 0 (normal state) to 15 (severe depression).

CONTACTS AND LOCATIONS:
Overall Officials: Henning Lohse-Busch, MD, Principal Investigator — Rheintalklinik
Locations (1):
- Rheintalklinik, Bad Krozingen, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No